CLINICAL TRIAL: NCT00293111
Title: An Open Label, Multi-Center, Phase II Study to Investigate the Safety and Efficacy of SDX-101 (R-Etodolac) in Patients With Relapsed or Refractory Multiple Myeloma (MM)
Brief Title: Safety and Efficacy of SDX-101 (R-Etodolac) in Patients With Relapsed or Refractory Multiple Myeloma (MM)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDX-101-04
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

INTERVENTIONS:
Drug: SDX-101 (R-Etodolac)

SUMMARY:
An Open Label, Multi-Center, Phase II Study to Investigate the Safety and Efficacy of SDX-101 (R-Etodolac) in Patients with Relapsed or Refractory Multiple Myeloma (MM)

ELIGIBILITY:
Inclusion Criteria:

1. Previously diagnosis of multiple myeloma as determined by any two of the major criteria, or major criteria 1 plus minor criteria b, c, or d, or major criteria 3 plus minor criteria a or c, or minor criteria a, b and c or a, b, and d.

   Major criteria:
   * Plasmacytomas on tissue biopsy
   * Bone marrow plasmacytomas (>30% plasma cells)
   * Monoclonal immunoglobulin spike on serum electrophoresis immunoglobulin G (IgG) >3.5 g/dl or immunoglobulin A (IGA) > 2.0 g/dl; kappa or lambda light chain excretion > 1 g/day on 24 hour urine protein electrophoresis

   Minor criteria:
   1. Bone marrow plasmacytomas (10 to 30% plasma cells)
   2. Monoclonal immunoglobulin present but of lesser magnitude than given under major criteria
   3. Lytic bone lesions
   4. Normal IgM < 50 mg/dl, IgA < 100 mg/dl, or IgG < 600 mg/dl
2. Has relapsed or refractory disease as determined by the following:

   Relapsed disease:

   • Disease progression developed following the achievement of at least stable disease or better to an anti-myeloma regimen.

   Refractory disease:

   • Disease progression developed during therapy with an anti-myeloma regimen prior to the achievement of at least stable disease or better. Includes the development of disease progression during maintenance or consolidation therapy with glucocorticoids or cytotoxic chemotherapy.
3. Age > 18 at signing of informed consent.
4. ECOG performance status 0-2.
5. Renal function 1.5 x upper limit normal (blood urea nitrogen [BUN], serum creatinine
6. Liver function ≤ 1.5 times upper limit of normal (total bilirubin, SGOT (AST) and SGPT (ALT) values).
7. Female patients of childbearing potential must have a negative pregnancy test (serum -human chorionic gonadotropin, -HCG); men and women of reproductive potential must employ effective contraceptive methods while on study therapy, and for 1 month following completion of treatment.
8. Signed IRB-approved informed consent by patient prior to all study related procedures.

Exclusion Criteria:

1. History of a prior malignancy with in the last 3 years with the exception of resected basal cell carcinoma, in situ cervical cancer at any time or other resected malignancies with no evidence of recurrence 5 or more years since diagnosis.
2. Patients with a hemoglobin count of < 8.0 g/dl, platelet count of < 50,000 cells/mm3, or an absolute neutrophil count (ANC) of < 1000 cells/mm3.
3. Serious infection, medical condition, or psychiatric condition that, in the opinion of the investigator, places the subject at unacceptable risk or might interfere with the achievement of the study objectives.
4. Chronic viral infection: positive hepatitis B or hepatitis C serology, known positive for human immunodeficiency virus (HIV) or human T-leukemia/lymphoma virus (HTLV).
5. Peptic ulcer disease (PUD) requiring treatment or surgical intervention within the last 2 years.
6. The use of steroids or chronic nonsteroidal anti-inflammatory drugs 28 days prior to the initiation of study medication.
7. Treatment with chemotherapy for the treatment of multiple myeloma or any investigational agent within 6 weeks of study entry.
8. History of allergy to NSAIDs or aspirin-induced asthma.
9. Pregnancy or currently breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-02; Primary Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas